CLINICAL TRIAL: NCT02947971
Title: Pilot Study for TCE (Tethered Capsule Endomicroscopy) Imaging of the Esophagus Using an OFDI (Optical Frequency Domain Imaging) Capsule With a Compact Imaging System
Brief Title: Pilot Study for TCE Imaging of the Esophagus Using an OFDI Capsule With a Compact Imaging System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-P000587; 5R01CA184102-02 (NIH)
Record Dates: First submitted 2016-04-14; First posted 2016-10-28 (Estimated); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Barrett's Esophagus
Keywords: Device; OFDI; Tethered Capsule Endomicroscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- OFDI Imaging (Experimental): Experimental OFDI Imaging
  Interventions: Device: Experimental OFDI Imaging

INTERVENTIONS:
Device: Experimental OFDI Imaging — Imaging of the esophagus with a compact OFDI system and distal scanning catheter

SUMMARY:
The goal of this research is to test a distal scanning capsule and a compact redesigned version of the OFDI imaging system in healthy and BE participants to assess ease of use, safety and feasibility in preparation for its use in a multicenter clinical trial.

DETAILED DESCRIPTION:
Ten healthy participants and ten participants with a previous diagnosis of Barrett's Esophagus (BE) will be enrolled in the study.

The capsule is attached to a string-like tether which allows the operator to control as well as navigate the capsule as it progresses down the esophagus using peristalsis.

Images of the esophagus will be acquired in real time to be analyzed later.

ELIGIBILITY:
Inclusion Criteria:

* A previous diagnosis of BE (not an inclusion criteria for healthy volunteers)
* Participants 18 years and older with a previous diagnosis of GERD
* Participants 14 years and older with a previous diagnosis of EoE (not an inclusion criteria for healthy volunteers)
* Health participants over the age of 18 but less than 85 years of age
* Participants must be able to give informed consent
* Participants must have no solid food for 4 hours prior to the procedure, and only clear liquids for 2 hours prior to the procedure.

Exclusion Criteria:

* Participants over 85 years of age
* Participants with the inability to swallow pills and capsules.
* Participants with a strong gag reflex
* Esophageal fistula and/or esophageal strictures with a stricture diameter that is smaller than the diameter of the capsule.
* Participants who are pregnant. In case of women of child bearing age, we will ask them if they are pregnant and if unsure; ask them to take a pregnancy test.

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-04-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of quality and performance of Compact Imaging System (CIS) | 5-7 Minutes of imaging
  Images obtained from the CIS will be assessed for quality and compared to images acquired from the previous imaging system

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No